CLINICAL TRIAL: NCT06144632
Title: Safety and Effectiveness Evaluation of the THERMOCOOL SMARTTOUCH SF Catheter With the TRUPULSE Generator for Treatment of Drug Refractory Symptomatic Paroxysmal Atrial Fibrillation (PAF)
Brief Title: A Study of the THERMOCOOL SMARTTOUCH Surround Flow (SF) Catheter With the TRUPULSE Generator for Treatment of Drug Refractory Symptomatic PAF
Acronym: SMARTPULSE PAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI202204; BWI202204 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2023-11-17; First posted 2023-11-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Drug Refractory Paroxysmal Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Group (Experimental): Participants with drug refractory, symptomatic paroxysmal atrial fibrillation will receive PFA /radiofrequency (RF) ablation using THERMOCOOL STSF catheter in conjunction with the TRUPULSE generator per the hospital's standard protocol (at discretion of investigator).
  Interventions: Device: THERMOCOOL STSF Bi- Directional Navigation Catheter; Device: TRUPULSE Generator

INTERVENTIONS:
Device: THERMOCOOL STSF Bi- Directional Navigation Catheter — THERMOCOOL STSF will be used in conjunction with TRUPULSE Generator to give pulsed field (PF) ablation or radiofrequency (RF) ablation.
Device: TRUPULSE Generator — TRUPULSE Generator will be used to deliver PF/RF ablation.

SUMMARY:
The purpose of this study is to demonstrate safety and effectiveness of the Biosense Webster (BWI) ablation system (THERMOCOOL SMARTTOUCH surround flow [STSF] catheter and TRUPULSE generator) when used for isolation of the atrial pulmonary veins (PVs) in treatment of participants with paroxysmal atrial fibrillation (PAF), an irregular heart rate that causing abnormal blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic paroxysmal atrial fibrillation (PAF) with (a) at least two symptomatic atrial fibrillation (AF) episodes within last six months from enrollment and (b) at least one AF episode electrocardiographically documented by electrocardiogram (ECG); transtelephonic monitoring (TTM), Holter monitor, telemetry strip or implanted device within 12 months prior to enrollment
* Failed at least one antiarrhythmic drug (AAD) (Class I or Class III) as evidenced by recurrent symptomatic AF, intolerable side effects to the AAD, or contraindication to the AAD
* Willing and capable of providing consent
* Able and willing to comply with all pre-, post- and follow-up testing and requirements

Exclusion Criteria:

* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause (for example, documented obstructive sleep apnea, acute alcohol toxicity, etcetera)
* Previously diagnosed with persistent AF (greater than [>] 7 days in duration)
* Previous left atrium (LA) ablation or surgery
* Participants known to require ablation outside the pulmonary vein (PV) region (for example, atrioventricular reentrant tachycardia, atrioventricular nodal reentry tachycardia, ventricular tachycardia, and Wolff-Parkinson-White), except cavotricuspid isthmus (CTI) lines for the ablation of typical right atrial flutter
* Documented severe dilatation of the LA (left anterior descending artery [LAD] >50mm) antero-posterior diameter on imaging within 6 months prior to enrollment
* Documented LA thrombus by imaging within 48 hours of the procedure
* Documented severely compromised left ventricular ejection fraction (LVEF less than [<] 40 percent [%]) by imaging within 6 months prior to enrollment
* Uncontrolled heart failure or New York Heart Association (NYHA) Class III or IV
* History of blood clotting, bleeding abnormalities or contraindication to anticoagulation (heparin) except subjects with prior left atrial appendage closure
* Documented thromboembolic event (including transient ischemic attack [TIA]) within the past 12 months
* Participants with unstable angina, percutaneous coronary intervention or acute myocardial infarction within 2 months
* Coronary artery bypass grafting (CABG) surgery within the past 6 months (180 days)
* Valvular cardiac surgical/percutaneous procedure (that is, ventriculotomy, atriotomy, valve repair or replacement and presence of a prosthetic valve)
* Unstable angina within 6 months
* Anticipated cardiac transplantation, cardiac surgery, or other major surgery within the next 12 months
* Significant pulmonary disease (for example, restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
* Significant congenital anomaly (for example, atrial septal defects [ASDs]) including repaired defects or medical problem that in the opinion of the investigator would preclude enrollment in this study
* Prior diagnosis of pulmonary vein stenosis
* Pre-existing hemi diaphragmatic paralysis
* Acute illness, active systemic infection, or sepsis
* Presence of intracardiac thrombus, myxoma, tumor, interatrial baffle or patch or other abnormality that precludes catheter introduction or manipulation
* Severe mitral regurgitation (Regurgitant volume greater than or equal to [>=] 60 milli liter (mL)/beat, Regurgitant fraction >= 50%, and/or Effective regurgitant orifice area >= 0.40 cm^2)
* Presence of implanted pacemaker, Implantable Cardioverter-Defibrillator (ICD), recently implanted (within 6 months) left atrial appendage occlusion (LAAO) device or other implanted metal cardiac device within cardiac space that may interfere with the energy field created during the ablation procedure
* Presence of a condition that precludes vascular access
* Current enrollment in an investigational study evaluating another device or drug
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal), lactating, or who are of child-bearing age and plan on becoming pregnant during the course of the clinical investigation
* Life expectancy less than 12 months
* Presenting contra-indications for the devices used in the study, as indicated in the respective Instructions for Use (IFU)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Primary Adverse Events (PAEs) | 7 days post-procedure
  PAEs occurring within 7 days of an ablation which uses the BWI ablation system (including atrio-esophageal fistula and pulmonary vein stenosis occurring greater than 7 days of post ablation procedure) will be reported.
Percentage of Participants with Freedom from Documented (Symptomatic and Asymptomatic) Atrial Fibrillation (AF), Atrial Tachycardia (AT), or Atrial Flutter (AFL) Episodes and Other Failure Modes | Up to 274 days
  The primary effectiveness endpoint for this study will be freedom from documented asymptomatic and symptomatic AF, AT, or AFL will be reported.

SECONDARY OUTCOMES:
Change From Baseline in Quality-of-Life (QOL) Improvement | From baseline to 12 months post ablation procedure
  Quality of life will be assessed as measured by the total Atrial Fibrillation Effect on Quality-of-Life (AFEQT) Questionnaire score. The score ranges from 0 to 100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster Inc. Clinical Trial, Study Director — Biosense Webster, Inc.
Locations (29):
- United States (29):
  - Grandview Medical Center, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Keck School of Medicine of USC, Los Angeles, California
  - HCA Florida JFK Hospital, Atlantis, Florida
  - Ascension St. Vincent's, Jacksonville, Florida
  - HCA Florida Mercy Hospital, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Georgia Arrhythmia Consultants and Research Institute, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - The Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Heart Specialist, Louisville, Kentucky
  - Massachusetts General, Boston, Massachusetts
  - Trinity Health Michigan Heart - Ann Arbor Campus, Ypsilanti, Michigan
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - NYU Langone Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Trident Medical Center, North Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor Scott & White Research Institute at The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Texsan, San Antonio, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Background] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society in Collaboration With the Society of Thoracic Surgeons. Circulation. 2019 Jul 9;140(2):e125-e151. doi: 10.1161/CIR.0000000000000665. Epub 2019 Jan 28. No abstract available. PMID 30686041
- [Background] Cain ME. Atrial fibrillation--rhythm or rate control. N Engl J Med. 2002 Dec 5;347(23):1822-3. doi: 10.1056/NEJMp020134. No abstract available. PMID 12466505
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Jackman WM, Wang XZ, Friday KJ, Roman CA, Moulton KP, Beckman KJ, McClelland JH, Twidale N, Hazlitt HA, Prior MI, et al. Catheter ablation of accessory atrioventricular pathways (Wolff-Parkinson-White syndrome) by radiofrequency current. N Engl J Med. 1991 Jun 6;324(23):1605-11. doi: 10.1056/NEJM199106063242301. PMID 2030716
- [Background] Jazayeri MR, Hempe SL, Sra JS, Dhala AA, Blanck Z, Deshpande SS, Avitall B, Krum DP, Gilbert CJ, Akhtar M. Selective transcatheter ablation of the fast and slow pathways using radiofrequency energy in patients with atrioventricular nodal reentrant tachycardia. Circulation. 1992 Apr;85(4):1318-28. doi: 10.1161/01.cir.85.4.1318. PMID 1555276
- [Background] Wilber DJ, Pappone C, Neuzil P, De Paola A, Marchlinski F, Natale A, Macle L, Daoud EG, Calkins H, Hall B, Reddy V, Augello G, Reynolds MR, Vinekar C, Liu CY, Berry SM, Berry DA; ThermoCool AF Trial Investigators. Comparison of antiarrhythmic drug therapy and radiofrequency catheter ablation in patients with paroxysmal atrial fibrillation: a randomized controlled trial. JAMA. 2010 Jan 27;303(4):333-40. doi: 10.1001/jama.2009.2029. PMID 20103757
- [Background] Marrouche NF, Dresing T, Cole C, Bash D, Saad E, Balaban K, Pavia SV, Schweikert R, Saliba W, Abdul-Karim A, Pisano E, Fanelli R, Tchou P, Natale A. Circular mapping and ablation of the pulmonary vein for treatment of atrial fibrillation: impact of different catheter technologies. J Am Coll Cardiol. 2002 Aug 7;40(3):464-74. doi: 10.1016/s0735-1097(02)01972-1. PMID 12142112
- [Background] Oral H, Knight BP, Tada H, Ozaydin M, Chugh A, Hassan S, Scharf C, Lai SW, Greenstein R, Pelosi F Jr, Strickberger SA, Morady F. Pulmonary vein isolation for paroxysmal and persistent atrial fibrillation. Circulation. 2002 Mar 5;105(9):1077-81. doi: 10.1161/hc0902.104712. PMID 11877358
- [Background] Pappone C, Oreto G, Rosanio S, Vicedomini G, Tocchi M, Gugliotta F, Salvati A, Dicandia C, Calabro MP, Mazzone P, Ficarra E, Di Gioia C, Gulletta S, Nardi S, Santinelli V, Benussi S, Alfieri O. Atrial electroanatomic remodeling after circumferential radiofrequency pulmonary vein ablation: efficacy of an anatomic approach in a large cohort of patients with atrial fibrillation. Circulation. 2001 Nov 20;104(21):2539-44. doi: 10.1161/hc4601.098517. PMID 11714647
- [Background] Haissaguerre M, Shah DC, Jais P, Hocini M, Yamane T, Deisenhofer I, Chauvin M, Garrigue S, Clementy J. Electrophysiological breakthroughs from the left atrium to the pulmonary veins. Circulation. 2000 Nov 14;102(20):2463-5. doi: 10.1161/01.cir.102.20.2463. PMID 11076817
- [Background] Duytschaever M, Vijgen J, De Potter T, Scherr D, Van Herendael H, Knecht S, Kobza R, Berte B, Sandgaard N, Albenque JP, Szeplaki G, Stevenhagen YJ, Taghji P, Wright M, Macours N, Gupta D. Standardized pulmonary vein isolation workflow to enclose veins with contiguous lesions: the multicentre VISTAX trial. Europace. 2020 Nov 1;22(11):1645-1652. doi: 10.1093/europace/euaa157. PMID 32879974
- [Background] Duytschaever M, De Pooter J, Demolder A, El Haddad M, Phlips T, Strisciuglio T, Debonnaire P, Wolf M, Vandekerckhove Y, Knecht S, Tavernier R. Long-term impact of catheter ablation on arrhythmia burden in low-risk patients with paroxysmal atrial fibrillation: The CLOSE to CURE study. Heart Rhythm. 2020 Apr;17(4):535-543. doi: 10.1016/j.hrthm.2019.11.004. Epub 2019 Nov 9. PMID 31707159
- [Background] Wojtaszczyk A, Caluori G, Pesl M, Melajova K, Starek Z. Irreversible electroporation ablation for atrial fibrillation. J Cardiovasc Electrophysiol. 2018 Apr;29(4):643-651. doi: 10.1111/jce.13454. Epub 2018 Mar 6. PMID 29399927
- [Background] Bohnen M, Stevenson WG, Tedrow UB, Michaud GF, John RM, Epstein LM, Albert CM, Koplan BA. Incidence and predictors of major complications from contemporary catheter ablation to treat cardiac arrhythmias. Heart Rhythm. 2011 Nov;8(11):1661-6. doi: 10.1016/j.hrthm.2011.05.017. Epub 2011 May 27. PMID 21699857
- [Background] Maor E, Sugrue A, Witt C, Vaidya VR, DeSimone CV, Asirvatham SJ, Kapa S. Pulsed electric fields for cardiac ablation and beyond: A state-of-the-art review. Heart Rhythm. 2019 Jul;16(7):1112-1120. doi: 10.1016/j.hrthm.2019.01.012. Epub 2019 Jan 11. PMID 30641148
- [Background] Zager Y, Kain D, Landa N, Leor J, Maor E. Optimization of Irreversible Electroporation Protocols for In-vivo Myocardial Decellularization. PLoS One. 2016 Nov 28;11(11):e0165475. doi: 10.1371/journal.pone.0165475. eCollection 2016. PMID 27893744
- [Background] Wittkampf FHM, van Es R, Neven K. Electroporation and its Relevance for Cardiac Catheter Ablation. JACC Clin Electrophysiol. 2018 Aug;4(8):977-986. doi: 10.1016/j.jacep.2018.06.005. Epub 2018 Jul 25. PMID 30139498
- [Background] Reddy VY, Neuzil P, Koruth JS, Petru J, Funosako M, Cochet H, Sediva L, Chovanec M, Dukkipati SR, Jais P. Pulsed Field Ablation for Pulmonary Vein Isolation in Atrial Fibrillation. J Am Coll Cardiol. 2019 Jul 23;74(3):315-326. doi: 10.1016/j.jacc.2019.04.021. Epub 2019 May 11. PMID 31085321
- [Background] Reddy VY, Koruth J, Jais P, Petru J, Timko F, Skalsky I, Hebeler R, Labrousse L, Barandon L, Kralovec S, Funosako M, Mannuva BB, Sediva L, Neuzil P. Ablation of Atrial Fibrillation With Pulsed Electric Fields: An Ultra-Rapid, Tissue-Selective Modality for Cardiac Ablation. JACC Clin Electrophysiol. 2018 Aug;4(8):987-995. doi: 10.1016/j.jacep.2018.04.005. Epub 2018 May 11. PMID 30139499
- [Background] Bardy GH, Coltorti F, Stewart RB, Greene HL, Ivey TD. Catheter-mediated electrical ablation: the relation between current and pulse width on voltage breakdown and shock-wave generation. Circ Res. 1988 Aug;63(2):409-14. doi: 10.1161/01.res.63.2.409. PMID 3396159
- [Background] DeSimone CV, Kapa S, Asirvatham SJ. Electroporation: past and future of catheter ablation. Circ Arrhythm Electrophysiol. 2014 Aug;7(4):573-5. doi: 10.1161/CIRCEP.114.001999. No abstract available. PMID 25140018
- [Background] van Driel VJ, Neven K, van Wessel H, Vink A, Doevendans PA, Wittkampf FH. Low vulnerability of the right phrenic nerve to electroporation ablation. Heart Rhythm. 2015 Aug;12(8):1838-44. doi: 10.1016/j.hrthm.2015.05.012. Epub 2015 May 18. PMID 25998897
- [Background] Schoellnast H, Monette S, Ezell PC, Deodhar A, Maybody M, Erinjeri JP, Stubblefield MD, Single GW Jr, Hamilton WC Jr, Solomon SB. Acute and subacute effects of irreversible electroporation on nerves: experimental study in a pig model. Radiology. 2011 Aug;260(2):421-7. doi: 10.1148/radiol.11103505. Epub 2011 Jun 3. PMID 21642418
- [Background] Tam AL, Abdelsalam ME, Gagea M, Ensor JE, Moussa M, Ahmed M, Goldberg SN, Dixon K, McWatters A, Miller JJ, Srimathveeravalli G, Solomon SB, Avritscher R, Wallace MJ, Gupta S. Irreversible electroporation of the lumbar vertebrae in a porcine model: is there clinical-pathologic evidence of neural toxicity? Radiology. 2014 Sep;272(3):709-19. doi: 10.1148/radiol.14132560. Epub 2014 Apr 25. PMID 24766034
- [Background] Li W, Fan Q, Ji Z, Qiu X, Li Z. The effects of irreversible electroporation (IRE) on nerves. PLoS One. 2011 Apr 14;6(4):e18831. doi: 10.1371/journal.pone.0018831. PMID 21533143
- [Background] Hong J, Stewart MT, Cheek DS, Francischelli DE, Kirchhof N. Cardiac ablation via electroporation. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:3381-4. doi: 10.1109/IEMBS.2009.5332816. PMID 19963798
- [Background] Reddy VY, Anter E, Rackauskas G, Peichl P, Koruth JS, Petru J, Funasako M, Minami K, Natale A, Jais P, Nakagawa H, Marinskis G, Aidietis A, Kautzner J, Neuzil P. Lattice-Tip Focal Ablation Catheter That Toggles Between Radiofrequency and Pulsed Field Energy to Treat Atrial Fibrillation: A First-in-Human Trial. Circ Arrhythm Electrophysiol. 2020 Jun;13(6):e008718. doi: 10.1161/CIRCEP.120.008718. Epub 2020 May 8. PMID 32383391
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412
- [Background] Reddy VY, Anic A, Koruth J, Petru J, Funasako M, Minami K, Breskovic T, Sikiric I, Dukkipati SR, Kawamura I, Neuzil P. Pulsed Field Ablation in Patients With Persistent Atrial Fibrillation. J Am Coll Cardiol. 2020 Sep 1;76(9):1068-1080. doi: 10.1016/j.jacc.2020.07.007. PMID 32854842
- [Background] Ekanem E, Reddy VY, Schmidt B, Reichlin T, Neven K, Metzner A, Hansen J, Blaauw Y, Maury P, Arentz T, Sommer P, Anic A, Anselme F, Boveda S, Deneke T, Willems S, van der Voort P, Tilz R, Funasako M, Scherr D, Wakili R, Steven D, Kautzner J, Vijgen J, Jais P, Petru J, Chun J, Roten L, Futing A, Rillig A, Mulder BA, Johannessen A, Rollin A, Lehrmann H, Sohns C, Jurisic Z, Savoure A, Combes S, Nentwich K, Gunawardene M, Ouss A, Kirstein B, Manninger M, Bohnen JE, Sultan A, Peichl P, Koopman P, Derval N, Turagam MK, Neuzil P; MANIFEST-PF Cooperative. Multi-national survey on the methods, efficacy, and safety on the post-approval clinical use of pulsed field ablation (MANIFEST-PF). Europace. 2022 Sep 1;24(8):1256-1266. doi: 10.1093/europace/euac050. PMID 35647644
- [Background] Gunawardene MA, Schaeffer BN, Jularic M, Eickholt C, Maurer T, Akbulak RO, Flindt M, Anwar O, Hartmann J, Willems S. Coronary Spasm During Pulsed Field Ablation of the Mitral Isthmus Line. JACC Clin Electrophysiol. 2021 Dec;7(12):1618-1620. doi: 10.1016/j.jacep.2021.08.016. Epub 2021 Sep 29. No abstract available. PMID 34600850
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation: Executive summary. J Arrhythm. 2017 Oct;33(5):369-409. doi: 10.1016/j.joa.2017.08.001. Epub 2017 Sep 15. No abstract available. PMID 29021841
- [Background] Chavez P, Messerli FH, Casso Dominguez A, Aziz EF, Sichrovsky T, Garcia D, Barrett CD, Danik S. Atrioesophageal fistula following ablation procedures for atrial fibrillation: systematic review of case reports. Open Heart. 2015 Sep 10;2(1):e000257. doi: 10.1136/openhrt-2015-000257. eCollection 2015. PMID 26380098
- [Background] Neven K, van Es R, van Driel V, van Wessel H, Fidder H, Vink A, Doevendans P, Wittkampf F. Acute and Long-Term Effects of Full-Power Electroporation Ablation Directly on the Porcine Esophagus. Circ Arrhythm Electrophysiol. 2017 May;10(5):e004672. doi: 10.1161/CIRCEP.116.004672. PMID 28487347
- [Background] Natale A, Reddy VY, Monir G, Wilber DJ, Lindsay BD, McElderry HT, Kantipudi C, Mansour MC, Melby DP, Packer DL, Nakagawa H, Zhang B, Stagg RB, Boo LM, Marchlinski FE. Paroxysmal AF catheter ablation with a contact force sensing catheter: results of the prospective, multicenter SMART-AF trial. J Am Coll Cardiol. 2014 Aug 19;64(7):647-56. doi: 10.1016/j.jacc.2014.04.072. PMID 25125294
- [Background] Reddy VY, Petru J, Funasako M, Kopriva K, Hala P, Chovanec M, Janotka M, Kralovec S, Neuzil P. Coronary Arterial Spasm During Pulsed Field Ablation to Treat Atrial Fibrillation. Circulation. 2022 Dec 13;146(24):1808-1819. doi: 10.1161/CIRCULATIONAHA.122.061497. Epub 2022 Sep 22. PMID 36134574
- [Background] Koruth JS, Dukkipati S, Carrillo RG, Coffey J, Teng J, Eby TB, Reddy VY, D'Avila A. Safety and efficacy of high-intensity focused ultrasound atop coronary arteries during epicardial catheter ablation. J Cardiovasc Electrophysiol. 2011 Nov;22(11):1274-80. doi: 10.1111/j.1540-8167.2011.02084.x. Epub 2011 Jun 15. PMID 21676047
- [Background] Ladejobi A, Christopoulos G, Tan N, Ladas TP, Tri J, van Zyl M, Yasin O, Sugrue A, Khabsa M, Uecker DR, Connolly RJ, Danitz DJ, DeSimone CV, Killu AM, Maor E, Holmes D, Asirvatham SJ, Del-Carpio Munoz F. Effects of Pulsed Electric Fields on the Coronary Arteries in Swine. Circ Arrhythm Electrophysiol. 2022 Oct;15(10):e010668. doi: 10.1161/CIRCEP.121.010668. Epub 2022 Oct 4. PMID 36194538
- [Background] Kovoor P, Ricciardello M, Collins L, Uther JB, Ross DL. Risk to patients from radiation associated with radiofrequency ablation for supraventricular tachycardia. Circulation. 1998 Oct 13;98(15):1534-40. doi: 10.1161/01.cir.98.15.1534. PMID 9769307
- [Background] Nahass GT. Fluoroscopy and the skin: implications for radiofrequency catheter ablation. Am J Cardiol. 1995 Jul 15;76(3):174-6. doi: 10.1016/s0002-9149(99)80053-8. No abstract available. PMID 7611155
- [Background] Calkins H, Niklason L, Sousa J, el-Atassi R, Langberg J, Morady F. Radiation exposure during radiofrequency catheter ablation of accessory atrioventricular connections. Circulation. 1991 Dec;84(6):2376-82. doi: 10.1161/01.cir.84.6.2376. PMID 1959193
- [Background] Lin, A.C. and D. Wilber, Complications associated with radiofrequency catheter ablation, in Radiofrequency Catheter Ablation of Cardiac Arrhythmias: Basic Concepts and Clinical Applications, S.K.S. Huang and D.J. Wilber, Editors. 2000, Futura Publishing Company, Inc.: Grouponk, NY. p. 737-746
- [Background] Scheinman MM, Huang S. The 1998 NASPE prospective catheter ablation registry. Pacing Clin Electrophysiol. 2000 Jun;23(6):1020-8. doi: 10.1111/j.1540-8159.2000.tb00891.x. PMID 10879389
- [Background] Cox B, Durieux ME, Marcus MA. Toxicity of local anaesthetics. Best Pract Res Clin Anaesthesiol. 2003 Mar;17(1):111-36. doi: 10.1053/bean.2003.0275. PMID 12751552
- [Background] Mertes PM, Laxenaire MC. Allergic reactions occurring during anaesthesia. Eur J Anaesthesiol. 2002 Apr;19(4):240-62. doi: 10.1017/s0265021502000418. PMID 12074414
- [Background] Morcos SK, Thomsen HS, Webb JA; Contrast Media Safety Committee of the European Society of Urogenital Radiology. Prevention of generalized reactions to contrast media: a consensus report and guidelines. Eur Radiol. 2001;11(9):1720-8. doi: 10.1007/s003300000778. PMID 11511894
- [Background] Gruchalla RS. 10. Drug allergy. J Allergy Clin Immunol. 2003 Feb;111(2 Suppl):S548-59. doi: 10.1067/mai.2003.93. PMID 12592301
- [Background] Bick RL, Frenkel EP. Clinical aspects of heparin-induced thrombocytopenia and thrombosis and other side effects of heparin therapy. Clin Appl Thromb Hemost. 1999 Oct;5 Suppl 1:S7-15. doi: 10.1177/10760296990050s103. PMID 10726030
- [Background] Thomson KR, Cheung W, Ellis SJ, Federman D, Kavnoudias H, Loader-Oliver D, Roberts S, Evans P, Ball C, Haydon A. Investigation of the safety of irreversible electroporation in humans. J Vasc Interv Radiol. 2011 May;22(5):611-21. doi: 10.1016/j.jvir.2010.12.014. Epub 2011 Mar 25. PMID 21439847
- [Background] Sugrue A, Vaidya VR, Livia C, Padmanabhan D, Abudan A, Isath A, Witt T, DeSimone CV, Stalboerger P, Kapa S, Asirvatham SJ, McLeod CJ. Feasibility of selective cardiac ventricular electroporation. PLoS One. 2020 Feb 21;15(2):e0229214. doi: 10.1371/journal.pone.0229214. eCollection 2020. PMID 32084220
- [Background] Cannon MJ, Goyne HE, Stone PJ, Macdonald LJ, James LE, Cobos E, Chiriva-Internati M. Modulation of p38 MAPK signaling enhances dendritic cell activation of human CD4+ Th17 responses to ovarian tumor antigen. Cancer Immunol Immunother. 2013 May;62(5):839-49. doi: 10.1007/s00262-013-1391-0. Epub 2013 Jan 25. PMID 23354626
- [Background] Deodhar A, Dickfeld T, Single GW, Hamilton WC Jr, Thornton RH, Sofocleous CT, Maybody M, Gonen M, Rubinsky B, Solomon SB. Irreversible electroporation near the heart: ventricular arrhythmias can be prevented with ECG synchronization. AJR Am J Roentgenol. 2011 Mar;196(3):W330-5. doi: 10.2214/AJR.10.4490. PMID 21343484
- [Background] Qin M, Liu X, Jiang WF, Wu SH, Zhang XD, Po S. Vagal response during pulmonary vein isolation: Re-recognized its characteristics and implications in lone paroxysmal atrial fibrillation. Int J Cardiol. 2016 May 15;211:7-13. doi: 10.1016/j.ijcard.2016.02.116. Epub 2016 Feb 23. PMID 26963618
- [Background] Yanagisawa S, Inden Y, Mizutani Y, Fujii A, Kamikubo Y, Kanzaki Y, Ando M, Funabiki J, Murase Y, Takenaka M, Otake N, Hattori T, Shibata R, Murohara T. Vagal response in cryoballoon ablation of atrial fibrillation and autonomic nervous system: Utility of epicardial adipose tissue location. J Arrhythm. 2017 Aug;33(4):275-282. doi: 10.1016/j.joa.2017.03.001. Epub 2017 Apr 24. PMID 28765757
- [Background] van Es R, Konings MK, Du Pre BC, Neven K, van Wessel H, van Driel VJHM, Westra AH, Doevendans PAF, Wittkampf FHM. High-frequency irreversible electroporation for cardiac ablation using an asymmetrical waveform. Biomed Eng Online. 2019 Jun 20;18(1):75. doi: 10.1186/s12938-019-0693-7. PMID 31221146
- [Background] Zupanic A, Ribaric S, Miklavcic D. Increasing the repetition frequency of electric pulse delivery reduces unpleasant sensations that occur in electrochemotherapy. Neoplasma. 2007;54(3):246-50. PMID 17447858
- [Background] Rombouts SJ, Nijkamp MW, van Dijck WP, Brosens LA, Konings M, van Hillegersberg R, Borel Rinkes IH, Hagendoorn J, Wittkampf FH, Molenaar IQ. Irreversible Electroporation of the Pancreas Using Parallel Plate Electrodes in a Porcine Model: A Feasibility Study. PLoS One. 2017 Jan 4;12(1):e0169396. doi: 10.1371/journal.pone.0169396. eCollection 2017. PMID 28052102
- [Background] Deshmukh A, Patel NJ, Pant S, Shah N, Chothani A, Mehta K, Grover P, Singh V, Vallurupalli S, Savani GT, Badheka A, Tuliani T, Dabhadkar K, Dibu G, Reddy YM, Sewani A, Kowalski M, Mitrani R, Paydak H, Viles-Gonzalez JF. In-hospital complications associated with catheter ablation of atrial fibrillation in the United States between 2000 and 2010: analysis of 93 801 procedures. Circulation. 2013 Nov 5;128(19):2104-12. doi: 10.1161/CIRCULATIONAHA.113.003862. Epub 2013 Sep 23. PMID 24061087
- [Background] Stewart MT, Haines DE, Verma A, Kirchhof N, Barka N, Grassl E, Howard B. Intracardiac pulsed field ablation: Proof of feasibility in a chronic porcine model. Heart Rhythm. 2019 May;16(5):754-764. doi: 10.1016/j.hrthm.2018.10.030. Epub 2018 Oct 30. PMID 30385383
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Sugrue A, Vaidya V, Witt C, DeSimone CV, Yasin O, Maor E, Killu AM, Kapa S, McLeod CJ, Miklavcic D, Asirvatham SJ. Irreversible electroporation for catheter-based cardiac ablation: a systematic review of the preclinical experience. J Interv Card Electrophysiol. 2019 Sep;55(3):251-265. doi: 10.1007/s10840-019-00574-3. Epub 2019 Jul 3. PMID 31270656
- [Background] Bradley CJ, Haines DE. Pulsed field ablation for pulmonary vein isolation in the treatment of atrial fibrillation. J Cardiovasc Electrophysiol. 2020 Aug;31(8):2136-2147. doi: 10.1111/jce.14414. Epub 2020 May 16. PMID 32107812
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Natale A, Albenque JP, Kautzner J, Shah D, Michaud G, Wharton M, Harari D, Mahapatra S, Lambert H, Mansour M. Randomized, Controlled Trial of the Safety and Effectiveness of a Contact Force-Sensing Irrigated Catheter for Ablation of Paroxysmal Atrial Fibrillation: Results of the TactiCath Contact Force Ablation Catheter Study for Atrial Fibrillation (TOCCASTAR) Study. Circulation. 2015 Sep 8;132(10):907-15. doi: 10.1161/CIRCULATIONAHA.114.014092. Epub 2015 Aug 10. PMID 26260733
- [Background] Cronin EM, Bogun FM, Maury P, Peichl P, Chen M, Namboodiri N, Aguinaga L, Leite LR, Al-Khatib SM, Anter E, Berruezo A, Callans DJ, Chung MK, Cuculich P, d'Avila A, Deal BJ, Della Bella P, Deneke T, Dickfeld TM, Hadid C, Haqqani HM, Kay GN, Latchamsetty R, Marchlinski F, Miller JM, Nogami A, Patel AR, Pathak RK, Saenz Morales LC, Santangeli P, Sapp JL Jr, Sarkozy A, Soejima K, Stevenson WG, Tedrow UB, Tzou WS, Varma N, Zeppenfeld K. 2019 HRS/EHRA/APHRS/LAHRS expert consensus statement on catheter ablation of ventricular arrhythmias. Heart Rhythm. 2020 Jan;17(1):e2-e154. doi: 10.1016/j.hrthm.2019.03.002. Epub 2019 May 10. PMID 31085023